CLINICAL TRIAL: NCT05601713
Title: Evaluating the Efficacy of Lower Leg Immersion With and Without Neck Cooling for Limiting Heat Strain in Elderly Adults During Extreme Heat Events
Brief Title: Mitigating Heat-induced Physiological Strain and Discomfort in Older Adults Via Lower Limb Immersion and Neck Cooling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University Research Chair, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-11-20-6234
Record Dates: First submitted 2022-10-19; First posted 2022-11-01 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Hyperthermia; Weather; Heat; Heat Stress; Heat Syncope; Aging
Keywords: Heat wave; Cooling intervention; Heat strain; Cardiovascular strain; Heat and health protection; Extreme heat events
MeSH Terms: conditions — Hyperthermia; Heat Stress Disorders

STUDY DESIGN:
Intervention Model Description: Participant will complete 3 simulated extreme heat event exposures in random order: i) no cooling intervention (control); ii) lower limb water immersion; and iii) lower limb water immersion with application of cool wet towel to the neck.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be informed of the study interventions before providing informed consent but will be masked to the specific trial until exposure (i.e., participants will not know the cooling intervention before the trial or during baseline measurements). Data will be blinded prior to analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No cooling intervention (control) (Active Comparator): Adults aged 65-85 years with or without type 2 diabetes and/or hypertension.
  Interventions: Other: No cooling (control)
- Lower limb immersion (Experimental): Adults aged 65-85 years with or without type 2 diabetes and/or hypertension.
  Interventions: Other: Lower limb immersion
- Lower limb immersion + neck cooling (Experimental): Adults aged 65-85 years with or without type 2 diabetes and/or hypertension.
  Interventions: Other: Lower limb immersion + neck cooling

INTERVENTIONS:
Other: No cooling (control) — Participants are exposed to 38°C, 35% relative humidity for 6 hours without cooling interventions (control condition). Drinking water is available ad libitum.
  Arms: No cooling intervention (control)
Other: Lower limb immersion — Participants are exposed to 38°C, 35% relative humidity for 6 hours. For the last 40 min of each hour, participants lower limbs are immersed in cool water (~20°C) up to the level of mid calf. Drinking water is available ad libitum.
  Arms: Lower limb immersion
Other: Lower limb immersion + neck cooling — Participants are exposed to 38°C, 35% relative humidity for 6 hours. For the last 40 min of each hour, participants lower limbs are immersed in cool water (~20°C) up to the level of mid calf. During limb immersion, a towel soaked in cool water (~20°C) is placed around the participants neck. The towel is re-wet half way through the 40-min limb immersion. Drinking water is available ad libitum.
  Arms: Lower limb immersion + neck cooling

SUMMARY:
The incidence and severity of hot weather and extreme heat events (heat waves) is increasing. As such, there is an urgent need to develop heat-alleviation strategies that can provide targeted protection for older adults who are at an elevated risk for heat-induced illnesses or death due to impaired body temperature and cardiovascular regulation. While air-conditioning provides the most effective protection from extreme heat, it is inaccessible for many individuals and cannot be used during power outages (e.g., heat-related rolling blackouts). Immersion of the lower limbs in cold water and/or the application of cold towels to the neck have been recommended as simple and sustainable alternatives to air-conditioning. However, empirical data to support the efficacy of these interventions for mitigating physiological strain and discomfort in older adults is lacking. To address this knowledge gap, this randomized crossover trial will evaluate the effect of lower limb immersion with and without application of cold towels to the neck on body core temperature, cardiovascular strain and autonomic function, dehydration, and thermal comfort in adults aged 65-85 years exposed to simulated heat wave conditions (38°C, 35% relative humidity) for 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults.
* Aged 65-85 years.
* Non-smoking.
* English or French speaking.
* Ability to provide informed consent.

Exclusion Criteria:

* Physical restriction (e.g., due to disease: intermittent claudication, renal impairment, active proliferative retinopathy, unstable cardiac or pulmonary disease, disabling stroke, severe arthritis, etc.).
* Use of or changes in medication judged by the patient or investigators to make participation in this study inadvisable (e.g., medications increasing risk of heat-related illness; beta blockers, anticholinergics, etc.)
* Cardiac abnormalities identified via 12-lead ECG during an incremental exercise test to volitional fatigue (performed for all participants).
* Peak aerobic capacity (VO2peak), as measured during an incremental exercise test to volitional fatigue, exceeding the 50th percentile of age- and sex-specific normative values published by the American College of Sports Medicine (ACSM).

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Core temperature | End of heat exposure (hour 6)
  Rectal temperature measured as an index of core temperature (15 minute average)

SECONDARY OUTCOMES:
Heart rate | End of heat exposure (hour 6)
  Heart rate derived from 3-lead electrocardiogram (15 minute average)
Systolic blood pressure | End of heat exposure (hour 6)
  Systolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures)
Diastolic blood pressure | End of heat exposure (hour 6)
  Diastolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures)
Rate pressure product | End of heat exposure (hour 6)
  Rate pressure product, an index of myocardial work and strain, calculated as systolic blood pressure x heart rate.
Heart rate variability: SDNN | End of heat exposure (hour 6)
  Standard deviation of normal-to-normal RR intervals (SDNN) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the seated position. SDNN will be evaluated twice, during two paced breathing periods (separated by 4 min of seated rest).
Heart rate variability: RMSSD | End of heat exposure (hour 6)
  Root mean squared standard deviation of normal-to-normal RR intervals (RMSSD) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the seated position. RMSSD will be evaluated twice, during two paced breathing periods (separated by 4 min of seated rest).
Cardiac response to standing from supine (30:15 ratio) | End of heat exposure (hour 6)
  Cardiac response to standing evaluated as the ratio between the highest RR interval (lowest heart rate) measured at the 30th heart beat after standing from supine (+/- 5 beats) and the lowest RR interval (highest heart rate) measured at the 15th heart beat after standing (+/- 5 beats). Cardiac response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest).
Systolic response to standing from supine | End of heat exposure (hour 6)
  Systolic blood pressure response to standing evaluated as the difference in blood pressure measured between the standing and supine. Standing systolic blood pressure will be taken as the lowest value of those measured after 60 and 120 seconds of standing. Systolic response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest).
Integrated baroreflex sensitivity (sit-to-stand maneuvers) | End of heat exposure (hour 6)
  Determined from beat-to-beat arterial pressures and heart rate (volume-clamp technique) during 5 min of sit-to-stand maneuvers performed at 0.05 Hz (3 cycles per min; 15 total cycles).
Fluid consumption | End of heat exposure (hour 6)
  Cumulative fluid consumption calculated by weighing participant water intake at the start and end of each hour of exposure.
Fluid loss | End of heat exposure (hour 6)
  Fluid loss calculated as the change in body mass during each exposure presented as a percentage of baseline body mass (corrected for food consumption)
Change in plasma volume | End of heat exposure (hour 6)
  Change in plasma volume from baseline values calculated from duplicate measurements of hemoglobin and hematocrit at the start and end of each exposure using the technique by Dill and Costill.
Thermal comfort | End of heat exposure (hour 6)
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") ranging from extremely uncomfortable to extremely comfortable (midpoint: neutral).
Orthostatic intolerance symptoms assessment | End of heat exposure (hour 6)
  Cumulative sum of scores on 6 questions asking participant to rank symptoms associated with orthostatic intolerance during the last 1-2 hours (including the lying-to-standing and sit-to-stand tests). All symptoms scored on a scale from 0 (none) to 10 (worst possible) and include feelings of: (1) "dizziness, lightheadedness, feeling faint, or feeling like you might black out"; (2) "Problems with vision (blurring, seeing spots, tunnel vision, etc.)"; (3) "Weakness"; (4) "Fatigue"; (5) "Trouble concentrating"; and (6) "Head and neck discomfort".

CONTACTS AND LOCATIONS:
Overall Officials: Glen P Kenny, PhD, Principal Investigator — University of Ottawa; Robert D Meade, PhD, Principal Investigator — University of Ottawa; Ronald J Sigal, MD, MPH, Principal Investigator — University of Calgary
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available with approved analysis plan and signed access agreement
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Following publication of the main study report(s)
Access Criteria: Approved analysis plan and signed access agreement